CLINICAL TRIAL: NCT05153915
Title: A Long-term, Open-label, Non-comparative Study to Evaluate the Safety and Efficacy of a Modigraf® Based Immunosuppression Regimen in De Novo Pediatric Allograft Liver and Kidney Transplantation Recipients
Brief Title: A Study to Evaluate the Safety and Efficacy of a Modigraf® Based Immunosuppression Regimen in De Novo Pediatric Allograft Liver and Kidney Transplantation Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F506-CL-0406; CTR20212679 (Registry Identifier: ChinaDrugTrials.org.cn); 2022-002351-19 (Registry Identifier: EudraCT)
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Liver Transplantation; Kidney Transplantation
Keywords: Liver Transplantation; Kidney Transplantation; Modigraf; Tacrolimus; Pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver Transplant (Experimental): Pediatric participants who undergo de novo allograft liver transplantation receive initial daily dose of 0.15 to 0.3 milligram per kilogram (mg/kg) of body weight oral suspension of tacrolimus granules post-operatively for 12 months.
  Interventions: Drug: Tacrolimus granules
- Kidney Transplant (Experimental): Pediatric participants who undergo de novo allograft kidney transplantation receive initial daily dose of 0.15 to 0.3 mg/kg of body weight oral suspension of tacrolimus granules post-operatively for 12 months.
  Interventions: Drug: Tacrolimus granules

INTERVENTIONS:
Drug: Tacrolimus granules — Oral
  Other Names: Modigraf
  Arms: Liver Transplant
Drug: Tacrolimus granules — Oral
  Other Names: Modigraf
  Arms: Kidney Transplant

SUMMARY:
The purpose of this study is to observe the safety and efficacy of Modigraf in de novo pediatric allograft liver and kidney transplantation recipients. This study will also monitor dose changes and tacrolimus whole blood trough levels of Modigraf based immunosuppression regimen.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent(s) or their legal representative(s), and participant where applicable agrees not to participate in another interventional study while participating in the present study from 1 month before screening to the end of the study.

Exclusion Criteria:

* Participant has previously received another organ transplant.
* Participant has a high immunological risk, defined as a panel reactive antibody (PRA) score > 50% in the previous 6 months (only applicable for kidney transplantation recipients).
* Cold ischemia time of the donor kidney longer than 30 hours (only applicable for kidney transplantation recipients).
* Bilateral kidney transplantation recipients (only applicable for kidney transplantation recipients).
* Participant receives an ABO incompatible donor organ.
* Participant has significant kidney impairment, defined as having serum creatinine ≥ 230 μmol/L (≥ 2.6 mg/dL) prior to transplantation (not applicable for kidney transplantation recipients).
* Participant has significant liver disease, defined as having elevated alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or total bilirubin (TBL) levels 3 times the upper value of the normal range prior to transplantation (not applicable for liver transplantation recipients).
* Participants with malignancies or a history of malignancy within the last 5 years.
* Participant has a significant, uncontrolled systemic infection and/or severe diarrhea, vomiting, active upper gastrointestinal disorder that may affect the absorption of tacrolimus or has an active peptic ulcer.
* Recipient or donor known to be human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) positive.
* Participant requires systemic immunosuppressive medication for any indication other than transplantation.
* Participants taking or requiring to be treated with medication or substances prohibited by this protocol.
* Known allergy or intolerance to steroids, macrolide antibiotics, basiliximab, or tacrolimus.
* Participants with severe primary disease/complications/poor general condition which may be unsuitable for participating in this study.
* Participant is currently participating in another clinical trial and/or has been taking any other study drug within 1 month prior to screening.
* Participant is unlikely to comply with the visits scheduled in the protocol.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Acute Rejection (AR) | From first dose to month 12
  AR is an immune response against the donor graft that causes tissue impairment and potential failure. The criteria for rejection was performed by the local histopathologist following the "Histological Grading of Liver Biopsies for Rejection", the "Banff diagnostic categories for renal allograft biopsies".
Percentage of Participants with Biopsy-Proven Acute Rejections (BPAR) | From first dose to month 12
  AR is an immune response against the donor graft that causes tissue impairment and potential failure. The criteria for rejection was performed by the local histopathologist following the "Histological Grading of Liver Biopsies for Rejection", the "Banff diagnostic categories for renal allograft biopsies". A BPAR episode was defined as any AR episode confirmed by biopsy.
Percentage of Participants with clinically suspected Rejection | From first dose to month 12
  AR is an immune response against the donor graft that causes tissue impairment and potential failure. The criteria for rejection was performed by the local histopathologist following the "Histological Grading of Liver Biopsies for Rejection", the "Banff diagnostic categories for renal allograft biopsies". An AR was clinically suspected in participants who experienced an increase in serum creatinine, after the exclusion of other causes of graft dysfunction (generally with biopsy).
Number of Participants who Died | From first dose to month 12
  Number of participants who died is recorded during 12 months' post-transplant; any cause of death was taken into account.
Number of participants with graft failure | From first dose to month 12
  Graft failure is defined as graft dysfunction including re-transplantation, graft loss or death, during the study period. A graft dysfunction to permanent dialysis in kidney transplantation was also considered as graft failure.
Number of dose adjustments throughout the study period | From first dose to month 12
  The number of dose changes will The dose adjustments required for the organ transplant were reported. The Safety Analysis Set (SAF) consisted of all participants who took at least one dose of study drug.
Number of participants with Treatment Emergent adverse events (AEs) | From first dose to month 12
  An AE is defined as any untoward medical occurrence in a participant administered a study drug not necessarily linked to this treatment. An AE can be any unfavorable and unintended sign (e.g., abnormal laboratory finding; abnormal laboratory test result or other safety assessment, symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug. Treatment emergent adverse event (TEAE) is defined as AE observed after administering the study drug.
Whole Blood Trough Levels of Tacrolimus | From month 1 through month 12 (predose)
  Tacrolimus whole blood trough levels are routinely monitored from whole blood samples, using a local assay method, for example EMITÒ or Liquid-Chromatography-Mass-Spectrometry-Mass-Spectrometry (LC-MS-MS) in the local laboratories.

CONTACTS AND LOCATIONS:
Overall Officials: Manager Medical Science, Study Director — Astellas Pharma China, Inc.
Locations (7):
- China (7):
  - Site CN86003, Beijing
  - Site CN86006, Changsha
  - Site CN86001, Guangzhou
  - Site CN86002, Shanghai
  - Site CN86007, Tianjin
  - Site CN86004, Wuhan
  - Site CN86005, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/F506-CL-0406/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26502&tenant=MT_AST_9011